CLINICAL TRIAL: NCT01290510
Title: Hyaluronan in the Treatment of Painful Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCHY106Tendon-2010-08
Record Dates: First submitted 2011-01-28; First posted 2011-02-07 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Tendinopathy
Keywords: tendinopathy; hyaluronan; tendon; hyaluronic acid
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hyaluronic acid sodium salt (Experimental)
  Interventions: Device: hyaluronic acid sodium salt

INTERVENTIONS:
Device: hyaluronic acid sodium salt — Two injections of 2 % (40 milligrams (mg) / 2 millilitres (ml)) hyaluronan in weekly interval.

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of TCHY106 (2% hyaluronan) in the treatment of painful tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 75 years of age and good general health condition.
* Signed written informed consent.
* Painful tendinopathy since ≥ 6 weeks.
* Pain according to Visual Analogue Scale (VAS; 100 millimetres (mm)) ≥ 40 mm.
* Ensured compliance of subjects for study period.

Exclusion Criteria:

* Treatment with any investigational product within 4 weeks prior to study entry.
* Patients with known hypersensitivity to the products (that is active compound and excipients) or any component or procedure used in the study.
* Severe intercurrent illness (for example: uncontrolled diabetes mellitus, peripheral neuropathy), which in the opinion of the investigator, may put the patient at risk when participating in the study, or affect the patient's ability to take part in the study.
* Concomitant disease at study relevant site influencing study evaluation.
* List of diseases or characteristics judged by the investigator to be incompatible with the assessments and/or procedures for the study evaluation.
* List of concomitant medications not allowed.
* Patients treated with: systemic and/or local steroids within the last 4 weeks, immunosuppressive drugs within the last 3 months, repeated use of non-steroidal anti-inflammatory drugs (NSAIDs) within the last week or occasional use within 24 hours.
* Recent history of drug and/or alcohol abuse (within the last 6 months).
* List of contra-indications to the treatment.
* Pregnant or lactating females.
* Fertile women who do not accept the consistent and correct use of highly effective methods of birth control defined as implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence or vasectomised partner during the treatment period and the first 4 weeks follow-up period.
* Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and or non completion of the study according to investigator's judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Visual Analogue Scale of pain (VAS; 100 millimetres (mm)) on day 35 | Baseline and Day 35

SECONDARY OUTCOMES:
Visual Analogue Scale of pain (VAS; 100 mm) on day 7 | On Day 7
Visual Analogue Scale of pain (VAS; 100 mm) on day 90 | On Day 90
Clinical parameters at baseline | At baseline
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical parameters on day 7 | On Day 7
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical parameters on day 35 | On Day 35
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical parameters on day 90 | On Day 90
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Quality of life questionnaire at baseline | At baseline
Quality of life questionnaire on day 7 | On Day 7
Quality of life questionnaire on day 35 | On Day 35
Quality of life questionnaire on day 90 | On Day 90
Patient's and investigator's global evaluation of study-relevant tendon complaints on day 7 | On Day 7
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition
Patient's and investigator's global evaluation of study-relevant tendon complaints on day 35 | On Day 35
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition
Patient's and investigator's global evaluation of study-relevant tendon complaints on day 90 | On Day 90
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition
Frequency of test product-related Adverse Events | Up to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Nils Lynen, Dr. med., Principal Investigator — Orthopädische Gemeinschaftspraxis Elisengalerie, Aachen (Germany)
Locations (2):
- Germany (2):
  - Zentrum für Orthopädie und Sportmedizin München, Munich, Bavaria
  - Orthopädische Gemeinschaftspraxis Elisengalerie, Aachen, North Rhine-Westphalia